CLINICAL TRIAL: NCT01291186
Title: The Effect of BMI on Median Effective Dose (ED50) of Intrathecal Hyperbaric Bupivacaine for Total Knee Replacement Arthroplasty
Brief Title: Effect of Body-mass Index (BMI) on Median Effective Dose of Intrathecal Hyperbaric Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul Medical Center (Other)
Responsible Party: Won Ho Kim M.D., Seoul Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SMC-2010-1-14
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-01

CONDITIONS: Arthroplasty, Knee
Keywords: spinal anesthesia; intrathecal bupivacaine; median effective dose; height
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- BPV6NO (Experimental)
  Interventions: Drug: BPV6NO
- BPV7NO (Experimental)
  Interventions: Drug: BPV7NO
- BPV8NO (Experimental)
  Interventions: Drug: BPV8NO
- BPV9NO (Experimental)
  Interventions: Drug: BPV9NO
- BPV10NO (Experimental)
  Interventions: Drug: BPV10NO
- BPV11NO (Experimental)
  Interventions: Drug: BPV11NO
- BPV6O (Active Comparator)
  Interventions: Drug: BPV6O
- BPV7O (Active Comparator)
  Interventions: Drug: BPV7O
- BPV8O (Active Comparator)
  Interventions: Drug: BPV8O
- BPV9O (Active Comparator)
  Interventions: Drug: BPV9O
- BPV10O (Active Comparator)
  Interventions: Drug: BPV10O
- BPV11O (Active Comparator)
  Interventions: Drug: BPV11O

INTERVENTIONS:
Drug: BPV6NO — intrathecal bupivacaine 6 mg for BMI less than 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV6NO
Drug: BPV7NO — intrathecal bupivacaine 7 mg for BMI less than 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV7NO
Drug: BPV8NO — intrathecal bupivacaine 8 mg for BMI less than 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV8NO
Drug: BPV9NO — intrathecal bupivacaine 9 mg for BMI less than 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV9NO
Drug: BPV10NO — intrathecal bupivacaine 10 mg for BMI less than 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV10NO
Drug: BPV11NO — intrathecal bupivacaine 11 mg for BMI less than 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV11NO
Drug: BPV6O — intrathecal bupivacaine 6 mg for BMI over 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV6O
Drug: BPV7O — intrathecal bupivacaine 7 mg for BMI over 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV7O
Drug: BPV8O — intrathecal bupivacaine 8 mg for BMI over 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV8O
Drug: BPV9O — intrathecal bupivacaine 9 mg for BMI over 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV9O
Drug: BPV10O — intrathecal bupivacaine 10 mg for BMI over 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV10O
Drug: BPV11O — intrathecal bupivacaine 11 mg for BMI over 27.5 kg/m2
  Other Names: bupivacaine; epinephrine
  Arms: BPV11O

SUMMARY:
The effect of Body-mass index (BMI) on requirements of local anesthetics used in spinal anesthesia has not been well established. The investigators tried to quantify the effect of BMI on spinal anesthesia by comparing the median effective dose of intrathecal bupivacaine between two different BMI groups.

DETAILED DESCRIPTION:
The effect of BMI on requirements of local anesthetics used in spinal anesthesia has not been well established. The investigators tried to quantify the effect of BMI on spinal anesthesia by comparing the median effective dose (ED50)of intrathecal bupivacaine between two different BMI groups. The investigators determined the ED50 and ED 95 of intrathecal hyperbaric bupivacaine of subjects with BMI below 27.5 kg/m2, and subjects with BMI over 27.5 kg/m2, respectively. By comparing the difference of ED50 and ED95 between the groups, the investigators tried to quantify the effect of BMI on the bupivacaine dose requirement.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective total knee replacement arthroplasty

Exclusion Criteria:

* Patients with previous spine surgery, diabetic and other neuropathy, skin infection at the site of injection, allergy to bupivacaine and other common contraindications for spinal anesthesia were excluded from this study.
* The patients with height less than 140 cm or more than 160 cm, body-mass index (BMI) less than 20 or greater than 35 were also excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
success of spinal anesthesia | every ten minutes during the surgery
  a bilateral T12 sensory level to pinprick within 10 min of the intrathecal drug administration with no additional epidural anesthetics required during the surgery

SECONDARY OUTCOMES:
time to first request for supplemental analgesia | every ten minutes during and after surgery
  for failure cases: it is the time of failure for success cases : it is the time of first postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, M.D., Principal Investigator — Seoul Medical Center
Locations (1):
- Seoul Medical Center, Seoul, South Korea